CLINICAL TRIAL: NCT04563247
Title: Seroprevalence of SARS-CoV 2 Among Asymptomatic Frontline Healthcare Workers During COVID 19: A Cross Sectional Study
Brief Title: Seroprevalence of SARS-CoV-2 in Asymptomatic Frontline COVID-19 HCWs
Status: Completed | Type: Observational
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Amina Asif, Assistant Professor, Lahore General Hospital
Other Study IDs: LGH002
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic frontline HCWs for COVID 19: All healthcare workers who worked in high exposure areas of hospital dealing with COVID 19.
  Interventions: Diagnostic Test: IgG SARS CoV 2 antibodies

INTERVENTIONS:
Diagnostic Test: IgG SARS CoV 2 antibodies — The asymptomatic healthcare workers of high exposure COVID19 areas will be tested for IgG SARS CoV 2 antibodies

SUMMARY:
This study is about the current knowledge on the immunological changes observed in various healthcare workers in this part of the world, who remained asymptomatic while working in high exposure areas of COVID-19 infection.

DETAILED DESCRIPTION:
Coronaviruses (CoVs) are enveloped, single positive-strand RNA viruses belonging to the large subfamily Coronavirinae, which can infect mammals and several other animals.The continued spread of coronavirus disease 2019 (COVID-19) has prompted widespread concern around the world, and the World Health Organization (WHO), on 11 March 2020, declared COVID-19 a pandemic. Studies on severe acute respiratory syndrome (SARS) and Middle East respiratory syndrome (MERS) showed that virus-specific antibodies were detectable in 80-100% of patients at 2 weeks after symptom onset. Currently, the antibody responses against SARS-CoV-2 remain poorly understood and the clinical utility of serological testing is unclear. Little is known about the kinetics, tissue distribution, cross-reactivity and neutralization antibody response in COVID-19 patients. Asymptomatic cases are common but to date there are scarce epidemiological surveys that provide a clear percentage of asymptomatic cases.

A large number of healthcare workers have been infected with the virus worldwide, presenting with severe symptoms to no symptoms at all, in which case being diagnosed on contact tracing only. The seropositivity rate in previously undiagnosed healthcare workers has been reported in different regions of the world. In a combined study of three hospitals of Turkey, the seropositivity rate of the previously undiagnosed HCWs was 2.7%. A study done in China revealed 17.5 % seropositivity rate.

This study will aim to comprehensively review the current knowledge on the immunological changes observed in various healthcare workers in this part of the world, who remained asymptomatic while working in high exposure areas of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* All HCWs who had been working in high exposure areas of COVID 19

Exclusion Criteria:

* Any HCW of high exposure areas of COVID 19 who suffered from COVID 19 themselves diagnosed on PCR or clinically

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Healthcare workers who have been working in high exposure areas of COVID 19 and havenot developed disease themselves while working in that area
Sampling Method: Probability Sample
Enrollment: 970 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
SARS CoV 2 IgG antibodies | 3 months
  The presence or absence of SARS CoV 2 antibodies in serum of HCWs

CONTACTS AND LOCATIONS:
Overall Officials: Amina Asif, MPhilMicro, Principal Investigator — LahoreGeneralHospital.Lahore
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided